CLINICAL TRIAL: NCT06908564
Title: Efficacy of BalancE RehabiliTation Based on Serious Games in People With Hip Arthroplasty: a Pilot Non-Randomized Multicenter Study
Brief Title: Balance Rehabilitation Based on Serious Games
Acronym: BERTHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP 23/08
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hip Replacement, Total
Keywords: Hip Arthroplasty Replacement; Lower Limb; Balance; Rehabilitation; Robotic-Assisted Therapy; Range Of Motion; Pain; Activity of Daily Living; Hip Replacement Total
MeSH Terms: conditions — Pain

STUDY DESIGN:
Masking Description: This study is assessor-blinded, meaning that the outcome assessors will be masked to group allocation to minimize bias in data collection and analysis. Other study personnel, including participants and intervention providers, will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (EG) (Experimental): The Experimental Group (EG) perform 30 minutes (16 sessions, 4 days/week, for 4 weeks) of balance rehabilitation exercises using non-immersive virtual reality with the OAK device (Khymeia Group, Italy).
  Interventions: Device: Experimental: Interactive balance rehabilitation based on serious games.
- Active comparator (CG) (Active Comparator): Partecipants assigned to Control Group (CG) follow 30 minutes (4 days/week, for 4 weeks) of conventional rehabilitative treatments for balance without the use of technological devices.
  Interventions: Other: Active Comparator: conventional balance rehabilitation without the use of technological devices.

INTERVENTIONS:
Device: Experimental: Interactive balance rehabilitation based on serious games. — The intervention of the Experimental Group consists of 30 minutes (16 sessions, 4 days/week, for 4 weeks) of balance rehabilitation exercises using non-immersive virtual reality through the OAK device (Khymeia Group, Italy). The system includes exercises that require the patient to reach visual targets by shifting their Center of Pressure (COP). The exercises are categorized based on the direction of COP displacement and can be performed with increasing difficulty, as determined by the physiotherapist during the rehabilitation process.
  Arms: Experimental Group (EG)
Other: Active Comparator: conventional balance rehabilitation without the use of technological devices. — Intervention of the Control Group (CG) consists of 30 minutes (4 days/week, for 4 weeks) of conventional balance rehabilitation treatments without the use of technological devices. The motor exercises will focus on the rehabilitation of balance, the trunk, and the lower limbs and will be carried out with a physiotherapist who will tailor the treatment according to the patient's characteristics and needs. Primary attention will be given to recovering trunk control and seated posture. This phase will focus on restoring and maintaining muscle trophism in the anterior and posterior kinetic chains of the thigh and lower leg, as well as the hip's range of motion, through isometric exercises and gentle joint mobilizations while adhering to anti-dislocation guidelines.
  The process will continue with the reacquisition of the upright stance, emphasizing proprioceptive, coordination, and balance abilities. Once the upright position is stabilized, gait re-education will be introduced.
  Arms: Active comparator (CG)

SUMMARY:
The effects of new technologies, particularly exergames, on the rehabilitation process of patients with hip arthroplasty have not yet been verified. For this reason, the aim of this study is to evaluate the effectiveness, in terms of balance recovery, of a balance rehabilitation program based on serious games in individuals with hip arthroplasty compared to conventional treatment.

DETAILED DESCRIPTION:
Total Hip Arthroplasty (THA) is one of the most commonly performed orthopedic surgeries worldwide, primarily aimed at reducing pain, improving function, and enhancing quality of life. Over the past decade, the rate of THA has increased by 30%, and it is projected to double by 2035. Rehabilitation after THA includes pain management, wound care, self-care, motor therapy, early mobilization, and complication prevention [iv, v, vi]. Active patient involvement in the rehabilitation process is increasingly recognized as essential for improving post-THA autonomy .

Exergames can enhance patient engagement and attention during treatment, potentially leading to better rehabilitation outcomes. The application of game design approaches in rehabilitation has gained popularity, offering more engaging treatments that boost patient motivation and understanding. Serious games, which are not primarily intended for entertainment, focus on specific therapeutic goals. In motor rehabilitation, exergames allow patients to perform physical exercises through video game interaction, often integrating sensors and biosensors that provide biofeedback and enable therapists to monitor progress and personalize treatment.

Despite their growing popularity, there is limited literature on the effectiveness and safety of exergames in orthopedic rehabilitation. A systematic review by Wang et al. found a moderate reduction in pain with technology-assisted rehabilitation (via tele-rehabilitation) in patients with hip and knee arthroplasty, but no significant effects on functional mobility. Research specifically on THA patients is scarce and of low quality. Byra et al. reported similar findings, indicating a lack of comprehensive evidence on the effectiveness of technological rehabilitation in THA patients, although preliminary results in pain management, posture training, and proprioception are promising.

The effects of new technologies, particularly exergames, on the rehabilitation of patients with hip arthroplasty remain unverified. This study aims to evaluate the effectiveness of a balance rehabilitation program based on serious games in individuals with hip arthroplasty compared to conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* First elective hip arthroplasty;
* Cognitive ability to understand and perform the exercises outlined in the protocol;
* Ability to sign the informed consent.

Exclusion Criteria:

* Unable to adhere to the exercise program due to poor compliance;
* Previous contralateral hip arthroplasty;
* Surgical wound complications;
* Severe cognitive, linguistic, or visual impairments (inability to understand and follow the study procedures);
* Conditions that, in the investigator's judgment, may interfere with the study or contraindicate participation for safety reasons;
* Diagnosis of epilepsy;
* Presence of implanted cardiac pacemakers;
* Lack of signed informed consent for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Time Up and Go Test (TUG) | Day 0 (T0 - baseline), day 30 (T1 - After treatment).
  Time up and go test assess fall risk and measure the progress of balance, sit to stand and walking.
  Simple screening test that is a sensitive and specific measure of probability for falls among older adults.
  This test is intended to population affected by Parkinson's Disease, Multiple Sclerosis, Alzheimer's, Hip fracture, Total Knee Arthroplasty, Total Hip Replacement, Stroke and Huntington Disease. Materials needed consist in one chair with armrest, stopwatch and tape for mark 3 meters. Patients wear their regular footwear and can use a walking aid, if needed.
  The patient starts in a seated position and stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down.
  The time stops when the patient is seated. Be sure to document the assistive device used. The score is calculated in seconds and high scores indicate an elevate risk of falling.

SECONDARY OUTCOMES:
Cognitive Time Up and Go Test (TUG-C) | Day 0 (T0 - baseline), day 30 (T1 - After treatment).
  Time up and go test assess fall risk and measure the progress of balance, sit to stand and walking. Simple screening test that is a sensitive and specific measure of probability for falls among older adults. Materials needed consist in one chair with armrest, stopwatch and tape for mark 3 meters. Patients wear their regular footwear and can use a walking aid, if needed. The patient starts in a seated position and stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down meanwhile he counting backwards in threes from a random start point. The time stops when the patient is seated. Be sure to document the assistive device used. The score is calculated in seconds and high scores indicate an elevate risk of fallTUG
Passive Range of Motion (p-ROM) | Day 0 (T0 - baseline), day 30 (T1 - After treatment).
  Passive ROM refers to the movement of a joint through its range of motion by an external force. It's calculated using goniometer. Goniometer measures with a sensitivity of 1 degree. Elevated degrees of p-rom means high joint mobility.
Ten Meter Walking Test (10MWT) | Day 0 (T0 - baseline), day 30 (T1 - After treatment).
  The 10 Metre Walk Test is a performance measure used to assess walking or gait speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function. Equipment required consists of a walkway of 10m with additional 2m at both ends, marked with tape, for acceleration & deceleration (14 m total). The 14-metre walkway is marked 0-, 2-, 12-, and 14-metre points. In addition is required 2 chairs and stopwatch (or timer). The total time taken to ambulate 10 meters is recorded in this way: timing starts when the toes pass the 2-meter mark and stops when the toes pass the 12-meter mark. The total time is recorded in m/s. Low total time in 10MWT means that gait speed is elevate.
Hip Dysfunction and Osteoarthritis Outcome Score for Joint Replacement (HOOS JR). | Day 0 (T0 - baseline), day 30 (T1 - After treatment).
  The hip disability and osteoarthritis outcome score (HOOS) is a questionnaire intended to be used to assess patient's opinions about their hip and associated problems and to evaluate their symptoms and functional limitations during a therapeutic process. HOOS JR is developed based on the original 40-question questionnaire HOOS. HOOS JR has 6 items and it is shorter than original HOOS.
  The HOOS is meant to be used over short and long-term intervals to assess changes over time or the effect of treatment. Factors that should be considered when using the HOOS include age, sex, weight, geographic location, other chronic diseases, history of an inactive hip problem, contralateral hip disease, and active knee, ankle, or foot problems. Each question allows for a score ranging from 0 to 4, where 0 corresponds to the absence of symptoms and 4 corresponds to the most severe symptom.
Medical Research Council Scale (MRC) | Day 0 (T0 - baseline), day 30 (T1 - After treatment).
  The Medical Research Council Scale (also known as Oxford Scale) is a numerical rating scale used to quantify the power or strength produced by the contraction of a muscle. The main muscle groups investigated are:
  Ankle Dorsiflexion, Ankle Plantiflexion, Knee Extension, Knee Flexion, Hip Flexion and Hip Extension. Muscle Grading Scores consists in:
  0-No detectable muscle contraction (visible or palpation);
  1. Detectable contraction (visible or palpation), but no movement achieved;
  2. Limb movement achieved, but unable to move against gravity;
  3. Limb movement against resistance of gravity;
  4. Limb movement against gravity and external resistance;
  5. Normal strength.
Modified Barthel Index (mBI) | Day 0 (T0 - baseline), day 30 (T1 - After treatment).
  The Barthel Index for Activities of Daily Living is an ordinal scale which measures a person's ability to complete activities of daily living (ADL). The Barthel Index measures the degree of assistance required by an individual on ten mobility and self-care ADL items. The ten items are scored with a number of points, and then a final score is calculated by summing the points awarded to each functional skill. This allows the examiner to measure a patient's functional disability by quantifying their performance. Scores can be assigned either via direct assessment / observation or from reliable interviews with the patient, family, or staff. Research also suggests that the examiner's "common sense" and clinical experience can be used to assign scores. The higher the score, the more independent the patient is in completing the measured ADLs. Higher scores also indicate the patient is more likely to return home, with varying degrees of assistance, following hospital discharge.
Visual Analog Scale (VAS) | Day 0 (T0 - baseline), day 30 (T1 - After treatment) and day 120 (T2 - 3 months after treatment).
  A Visual Analogue Scale (VAS) is one of the pain rating scales.It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. From the patient's perspective, this spectrum appears continuous; their pain does not take discrete jumps, as a categorization of none, mild, moderate and severe would suggest. It was to capture this idea of an underlying continuum that the VAS was devised. The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions.
  The VAS allows you to assign a value to pain from 1 to 10, where 1 corresponds to no pain and 10 corresponds to the maximum pain perceived by the patient in his life.
Activities-specific Balance Confidence scale (ABC). | Day 0 (T0 - baseline), day 30 (T1 - After treatment) and day 120 (T2 - 3 Months after treatment).
  Activities-specific balance confidence (ABC) scale is a structured questionnaire that measures an individual's confidence during ambulatory activities without falling or experiencing a sense of unsteadiness. It consists of 16 questions gauging the individual's confidence while doing activities. The ABC scale is reported to be an accurate measure to identify individuals with a fall risk in populations of stroke, multiple sclerosis, Parkinson's, vestibular disorders, in elderly, and in other neurological conditions that can affect balance. Its a 16-item questionnaire where patients' rate their confidence while doing activities with a scoring from 0-100 (0 is no confidence and 100 is full confidence).

OTHER OUTCOMES:
Bilateral thigh cytometry. | Day 0 (T0 - baseline), day 30 (T1 - After treatment).
  The measurement of the thigh circumference is performed on both legs. The measurement is taken at the root of the thigh, approximately 1 cm below the gluteal fold.
Number of falls in the last 3 months. | Day 0 (T0 - baseline), day 30 (T1 - After treatment) and day 120 (T2 - 3 months after treatment).
  The circumference of the thigh of both legs is measured. The measurement is taken at the root of the thigh, that is, approximately 1 cm below the gluteal fold.
Client satisfaction questionnaire . | Day 30 (T1 - After treatment).
  The Client satisfaction questionnaire investigates the subject's overall satisfaction with participating in the study. It consists of six questions with a score ranging from 0 to 4. A high score corresponds to a high level of satisfaction from the subject.
Posturography | Day 0 (T0 - baseline), day 30 (T1 - After treatment).
  Posturography (or stabilometry) is an examination that allows for the assessment and measurement of fine postural control. The examined subject stands on a computerized and sensorized platform, remaining still in an upright position. The recording lasts 30 seconds and is repeated twice with eyes open and arms at the sides, and twice with eyes closed and arms at the sides.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Marco Franceschini, MD, Study Chair — IRCCS San Raffaele Roma; Prof. Marco Franceschini, MD, Principal Investigator — IRCCS San Raffaele Roma
Locations (2):
- Italy (2):
  - IRCCS San Raffaele Roma, Rome, Italy
  - Casa di Cura San Raffaele Sulmona, Sulmona, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcome measures will be shared, including assessment results and relevant demographic data, in compliance with ethical and legal requirements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available after official publication and upon request.
Access Criteria: Access will be granted upon specific request to the Study Chair, Principal Investigator, Sub-Investigator, or Central Study Contact Person. Researchers must submit a formal proposal outlining the intended use of the data, which will be reviewed for scientific merit and ethical compliance. Approved requests will receive access through a secure data-sharing platform.